CLINICAL TRIAL: NCT01286233
Title: Biobehavioral Mechanisms of Fatigue in Patients Treated on NCIC CTG MA.32: A Phase III Randomized Trial of Metformin Versus Placebo on Recurrence and Survival in Early Stage Breast Cancer
Brief Title: Study of Biomarkers Associated With Fatigue in Patients With Early-Stage Breast Cancer Treated With Metformin or Placebo on NCIC-CTG-MA.32
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP MA.32.F; NSABP-NCIC-CTG-MA.32.F
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Depression; Fatigue; Sleep Disorders
Keywords: fatigue; sleep disorders; depression; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Sleep Wake Disorders | interventions — Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Metformin: 850 mg orally twice a day for 5 years
  Interventions: Drug: Metformin
- Group 2: Placebo: One caplet orally twice a day for 5 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin
  Groups: Group 1: Metformin
Drug: Placebo
  Groups: Group 2: Placebo

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with breast cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to fatigue.

PURPOSE: This research study is studying biomarkers associated with fatigue in patients with early-stage breast cancer treated with metformin or placebo on NCIC-CTG-MA.32.

DETAILED DESCRIPTION:
OBJECTIVES:

* To prepare, separate into components, and store the blood specimens at the NSABP Serum Bank at Baylor College of Medicine Breast Center for future DNA, RNA, and plasma analysis, and to analyze specific proinflammatory cytokines, genetic polymorphisms, and RNA expression arrays in collaborating laboratories at University of California, Los Angeles (UCLA).
* To examine the association between markers of inflammation and symptoms of fatigue among patients with and without exposure to metformin hydrochloride.
* To examine the relationship between single nucleotide polymorphism (SNPs) in the promoter regions of IL-1 and IL-6 and symptoms of fatigue with and without exposure to metformin hydrochloride.
* To examine RNA expression profiles in relationship to fatigue and compare the pattern of expression in patients with and without exposure to metformin hydrochloride.
* To determine the biological and behavioral predictors of fatigue in breast cancer patients in the five years post-randomization.
* To determine whether metformin is associated with reductions in inflammatory markers and corresponding decreases in fatigue. (Exploratory)

OUTLINE: This is a multicenter study.

Patients' serum and plasma, collected at baseline and at 6, 12, and 24 months after NCIC CTG MA.32 randomization, are analyzed for inflammatory markers, DNA polymorphisms, and RNA expression arrays by ELISA, TaqMan PCR, and RT-PCR.

Patients complete the Fatigue Symptom Inventory (symptoms associated with fatigue, sleep disturbance, depression, and endocrine therapy) at baseline and periodically during study.

ELIGIBILITY:
Inclusion Criteria

* The patient must have consented to participate and must have signed and dated an appropriate IRB-approved consent form that conforms to federal and institutional guidelines for the MA.32.F Study before being enrolled.
* The patient must be female.
* The patient must reside in the United States or Canada.
* The patient must be English-speaking.
* The patient must be eligible for randomization in the MA.32 treatment trial. (Participation in the MA.32 QOL study is permitted but not required.)
* The patient must not have started taking MA.32 study therapy.
* The patient must have completed primary breast radiation therapy at least two weeks prior to enrollment in MA.32.F.

Exclusion Criteria

* MA.32 study therapy has been initiated.
* Currently receiving radiation therapy or additional radiation therapy is planned for initiation after starting MA.32 study therapy.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who have been diagnosed and have undergone definitive surgical treatment for invasive breast cancer within the previous 12 months and who are eligible for randomization to NCIC MA.32.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2011-07; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Questionnaire scores from patient reported outcome battery regarding fatigue, stress, sleep, depression, and general quality of life | Collected at baseline and 6, 12, 24, and 36 months from randomization
Questionnaire scores from patient reported comorbid conditions and behavioral risks | Collected at baseline and 6, 12, 24, and 36 months from randomization
Biological correlates of fatigue (medical and demographic characteristics of pts.) | Collected at baseline and 6, 12, 24, and 36 months from randomization
  Biological correlates (medical) will be collected at these timepoints. Standard demographics will be collected at baseline only.
DNA polymorphisms | Collected at baseline
Changes in RNA gene expression | Collected at baseline and 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (256):
- United States (252):
  - Kaiser Permanente Medical Center - Anaheim/Orange County, Anaheim, California
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente Medical Center - Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - Kaiser Permanente Medical Center - Fontana, Fontana, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Harbor City, Harbor City, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente - Irvine, Irvine, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Kaiser Foundation Hospital - West Los Angeles, Los Angeles, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente - Ontario Vineyard Medical Offices and Ambulatory SurgiCenter, Ontario, California
  - Kaiser Permanente Medical Group, Panorama City, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Riverside, Riverside, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Medical Cener - Woodland Hills, Woodland Hills, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
- Canada (4):
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - St. Catharines General Hospital at Niagara Health System, Saint Catharines, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario